CLINICAL TRIAL: NCT06912672
Title: Performance Evaluation of a Urine-based Methylation Assay for Urothelial Carcinoma in Patients With Hematuria: A Prospective, Multi-center Cohort Study
Brief Title: Performance Evaluation of a Urine-based Methylation Assay for Urothelial Carcinoma
Acronym: UMT-UC
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Epiprobe Biotechnology Co., Ltd. (Industry)
Collaborators: Changhai Hospital (Other); RenJi Hospital (Other); Tongji Hospital (Other); First Hospital of China Medical University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: EPI-UC-2025-01
Record Dates: First submitted 2025-04-02; First posted 2025-04-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial Carcinoma; Hematuria; DNA methylation
MeSH Terms: conditions — Carcinoma, Transitional Cell; Hematuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Urine sediment DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Evaluate the diagnostic performance of EPIPROBE TAGMe DNA Methylation Detection Kit for Urothelial Cancer — The study aims to evaluate the diagnostic performance of the EPIPROBE TAGMe DNA Methylation Detection Kit for the detection of urothelial cancer. This assay utilizes targeted DNA methylation analysis to identify specific epigenetic alterations associated with urothelial malignancies. The performance of the kit will be assessed in terms of sensitivity, specificity, and overall diagnostic accuracy using clinical urine samples from a patient population with hematuria.

SUMMARY:
Urothelial carcinoma (UC) is the most common malignancy of the urinary system. Hematuria is a significant clinical manifestation of UC, often diagnosed through invasive procedures. Urine DNA methylation testing is a promising non-invasive method for early UC detection. To evaluate the sensitivity and specificity of urine DNA methylation testing for detecting UC, using standard clinical and pathological diagnoses as the gold standard.

DETAILED DESCRIPTION:
Urothelial carcinoma (UC) is the most common malignancy of the urinary system, and early detection and diagnosis are crucial for patient prognosis. Hematuria is a significant clinical manifestation of UC, but its diagnosis often relies on invasive procedures and imaging, posing a substantial burden on patients. With the advancement of molecular biology techniques, urine DNA methylation testing has emerged as a non-invasive and highly sensitive method for early UC detection. This study aims to evaluate the performance of urine DNA methylation testing in detecting UC in patients with hematuria.

All patients with hematuria will receive standard clinical diagnosis, including examinations, tests, surgeries, and pathological assessments to determine the presence of UC. These clinical diagnoses will serve as the gold standard to evaluate the sensitivity and specificity of urine DNA methylation testing in detecting UC in patients with hematuria.

To ensure accuracy and reliability of the results, select a subset of samples with known test results for external methylation sequencing. Authorized researchers will unblind the samples, and the statistical team will analyze the results, calculating sensitivity, specificity, positive predictive value, and negative predictive value of the urine DNA methylation test.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 90 years, with gross or microscopic hematuria.
* Able to provide enough urine for testing before surgery.
* Consent to participate in the study and sign the informed consent form.

Exclusion Criteria:

* With history of any malignancies (including Urothelial carcinoma).
* Severe urinary tract infection leading to sepsis.
* Patients with indwelling catheters, nephrostomy, or cystostomy.
* Severe liver or kidney failure or other conditions deemed unsuitable for the study.
* Samples with insufficient DNA content or other quality control failures.
* Incomplete clinical or pathological data.
* Patients currently undergoing intravesical or systemic chemotherapy, radiotherapy, immunotherapy, or targeted therapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The initial population suspected of having urothelial carcinoma with hematuria
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of DNA methylation test for urothelial carcinoma | 2 weeks
  Evaluate the diagnostic performance of EPIPROBE TAGMe DNA Methylation Detection Kit for Urothelial Cancer by calculating the sensitivity, specificity.

IPD SHARING:
Plan to Share IPD: No